CLINICAL TRIAL: NCT04535986
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Ensifentrine Over 24 Weeks (With a 48-week Safety Subset) in Subjects With Moderate to Severe COPD
Brief Title: A Phase 3 Clinical Trial to Evaluate the Safety and Efficacy of Ensifentrine in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPL554-CO-301
Record Dates: First submitted 2020-08-19; First posted 2020-09-02 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Ensifentrine Nebulized Suspension; 3 mg BID
  Interventions: Drug: Ensifentrine
- Arm 2 (Placebo Comparator): Placebo Nebulized BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ensifentrine — Dosage Formulation: Ensifentrine Nebulizer suspension Dosage 3mg Frequency: Twice Daily for 24 weeks or 48 weeks
  Arms: Arm 1
Drug: Placebo — Dosage Formulation: Ensifentrine Placebo Nebulizer solution Frequency: Twice Daily for 24 weeks or 48 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ensifentrine in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

Informed Consent

1. Capable of giving informed consent indicating that they understand the purpose of the study and study procedures and agree to comply with the requirements and restrictions listed in the informed consent form (ICF).

   Age and Sex
2. Age: Patient must be 40 to 80 years of age inclusive, at the time of Screening.
3. Sex:

   * Males are eligible to participate if they agree to use contraception as described in the contraceptive guidance from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication.
   * Females are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions apply:

     1. Not a woman of childbearing potential (WOCBP) as defined in Or
     2. A WOCBP who agrees to follow the contraceptive guidance from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication.

   Smoking History
4. Smoking History: Current or former cigarette smokers with a history of cigarette smoking ≥10 pack years at Screening (Visit 0) [number of pack years = (number of cigarettes per day / 20) × number of years smoked (eg, 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Pipe and/or cigar use cannot be used to calculate pack-year history. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 0. Smoking cessation programs are permitted during the study.

   COPD Diagnosis, Symptoms, Severity and Maintenance Therapy
5. COPD Diagnosis: Patients with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines with symptoms compatible with COPD.
6. COPD Symptoms: A score of ≥2 on the Modified Medical Research Council (mMRC) Dyspnea Scale.
7. COPD Severity:

   1. Pre- and Post-albuterol/salbutamol FEV1/FVC ratio of <0.70.
   2. Post-albuterol/salbutamol FEV1 ≥30 % and ≤70% of predicted normal calculated using the National Health and Nutrition Examination Survey III.
8. Maintenance Therapy: Patients on no maintenance/background therapy or patients on stable maintenance LAMA or LABA therapy are eligible. Patients taking maintenance LAMA or LABA therapy must demonstrate stable use of the maintenance LAMA or LABA therapy for at least 3 months prior to Screening and agree to continue use for the duration of the study. Background maintenance LAMA or LABA bronchodilator therapy will be capped at 50% of patients.

   Other Requirements for Inclusion
9. Capable of withholding SABAs for 4 hours prior to initiation of any spirometry. Patients in the maintenance LAMA or LABA therapy stratum must be capable of withholding Twice-Daily maintenance LAMA or LABA for 24 hours and Once-Daily maintenance LAMA or LABA for 48 hours prior to initiation of any spirometry.
10. Capable of using the study nebulizer correctly and complying with all study restrictions and procedures.
11. Ability to perform acceptable spirometry in accordance with ATS/ERS guidelines.

Inclusion Criteria at Randomization (RPL554-CO-301)

1. Symptoms of COPD: A score of ≥2 on the mMRC Dyspnea Scale.
2. Completion of the e-Diary at least 5 of the last 7 days of the Run-in period.

Exclusion Criteria:

Current Condition or Medical History

1. History of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
2. Hospitalizations for COPD, pneumonia, or Corona Virus Disease 2019 (COVID-19) in the 12 weeks prior to Screening and/or a positive COVID-19 test result indicating an active infection at Screening. Patients with COVID-19 antibodies from a previous exposure with no active infection are not excluded.
3. COPD exacerbation requiring oral or parenteral steroids within 3 months of Screening.
4. Previous lung resection or lung reduction surgery within 1-year of Screening.
5. Long term oxygen use defined as oxygen therapy prescribed for greater than 12 hours per day. As needed oxygen use (≤12 hours per day) is not exclusionary.
6. Pulmonary rehabilitation, unless such treatment has been in a stable maintenance phase for 4 weeks prior to Visit 1 and remains stable during the study.
7. Lower respiratory tract infection within 6 weeks of Screening.
8. Other respiratory disorders including, but not limited to, a current diagnosis of asthma, active tuberculosis, lung cancer, sarcoidosis, lung fibrosis, interstitial lung diseases, unstable sleep apnea, known alpha-1 antitrypsin deficiency, core pulmonale, clinically significant pulmonary hypertension, clinically significant bronchiectasis, or other active pulmonary diseases.
9. Major surgery (requiring general anesthesia) in the 6 weeks prior to Screening, lack of full recovery from surgery at Screening, or planned surgery through the end of the study.
10. Historical or current evidence of clinically significant cardiovascular disease defined as any disease that in the opinion of the Investigator would put the safety of the patient at risk through participation or which could affect the efficacy or safety analysis if the disease/condition were to exacerbate during the study, including, but not limited to:

    * Myocardial infarction or unstable angina within 6 months prior to Screening.
    * Unstable or life-threatening cardiac arrhythmia requiring intervention within 3 months prior to Screening.
    * Diagnosis of New York Heart Association Class III and Class IV heart failure.
11. Chronic uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric, or ophthalmic diseases that the Investigator believes are clinically significant.
12. Unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
13. History of or current malignancy of any organ system, treated or untreated within the past 5 years, except for localized basal or squamous cell carcinoma of the skin.
14. Findings on physical examination that an investigator considers to be clinically significant at Screening.

    Prior/Concomitant Therapy
15. Use of prohibited medications within the time intervals.

    History or Suspicion of Drug or Alcohol Abuse
16. Current or history of past drug or alcohol abuse within the past 5 years.

    Laboratory and Other Diagnostic Parameters
17. Glomerular Filtration Rate (eGFR) <30 mL/min. The Chronic Kidney Disease Epidemiology Collaboration Creatinine (2009) calculation will be used (Levey, 2009).
18. Alanine aminotransferase (ALT) ≥ 2 x upper limit of normal (ULN), alkaline phosphatase and/or bilirubin > 1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
19. Any other abnormal hematology, biochemistry, or viral serology deemed by an investigator to be clinically significantly abnormal. Abnormal chemistry and/or hematology may be repeated during Screening.
20. Chest X-ray (CXR; posterior-anterior) at Screening, or in the 12 months prior to Screening with clinically significant abnormalities not attributable to COPD. If a CXR within the past 12 months is not available but a computerized tomography (CT) scan within the same time period is available, the CT scan may be reviewed in place of a CXR. For subjects in Germany, if a CXR or CT scan is not available in the 12 months prior to Screening, the subject is not eligible for the study.
21. Electrocardiogram (ECG) finding that is significantly abnormal on the 12-lead ECG obtained at Screening.

    Other Exclusions
22. Use of an experimental drug within 30 days or 5 half-lives of Screening, whichever is longer, and/or participation in a study treatment-free follow-up phase of a clinical study within 30 days prior to Screening.
23. Use of an experimental medical device or participation in a follow-up phase of an experimental medical device clinical study within 30 days prior to Screening.
24. Intolerance or hypersensitivity to albuterol/salbutamol or ensifentrine (RPL554) or any of its excipients/components.
25. Prior receipt of blinded study medication in an ensifentrine (RPL554) study.
26. Affiliation with the investigator site, including an Investigator, Sub-Investigator, study coordinator, study nurse, other employee of participating investigator or study site or a family member of the aforementioned.
27. Inability to read, understand, and/or complete questionnaires (in the opinion of the Investigator).
28. A disclosed history or one known to the Investigator of significant non-compliance in previous investigational studies or with prescribed medications.
29. Any other reason that the Investigator considers makes the patient unsuitable to participate.

Exclusion Criteria at Randomization (RPL554-CO-301)

1. COPD exacerbation or lower respiratory tract infection between Screening and Randomization (defined as use of any additional treatment other than current treatment and rescue medication and/or emergency department or hospital visit). Patients with a severe COPD exacerbation that requires hospitalization may not be rescreened.
2. Positive COVID-19 result at Screening or between Screening and Randomization.
3. Prohibited medication use between Screening Visit 0 and Visit 1.
4. Significantly abnormal ECG finding on the 12-lead ECG obtained at Screening as assessed by the investigator or site medical doctor/medically qualified person or on the pre-dose (prior to randomization) ECG obtained at Visit 1.

   In the event that the central ECG reviewer discovers a significant ECG abnormality on the Visit 1 ECG, the patient will be discontinued.
5. Did not meet one or more of the Inclusion Criteria or met one or more of the Exclusion Criteria.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (121):
- United States (39):
  - Phoenix Medical Group, Peoria, Arizona
  - AMR Tempe, Tempe, Arizona
  - Beach Physicians Medical Group, Huntington Beach, California
  - Downtown LA Research Center, Inc., Los Angeles, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Qway Research, LLC, Hialeah, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Elite Clinical Research, Miami, Florida
  - Global Research Solutions Corp, Miami, Florida
  - Phoenix Medical Research, Miami, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - IACT Health, Rincon, Georgia
  - In-Quest Medical Research, LLC, Suwanee, Georgia
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Pulmonary Research Institute of SE Michigan, Farmington Hills, Michigan
  - Midwest Chest Consultants, Saint Charles, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Sierra Clinical Research, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - IMA Clinical Research, LLC, New York, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Remington Davis Clinical Research, Columbus, Ohio
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Clinical Research Associates of Central PA, LLC, DuBois, Pennsylvania
  - University of Pittsburgh Physicians, Emphysema/COPD Research Center, Pittsburgh, Pennsylvania
  - Medtrial, Columbia, South Carolina
  - MDFirst Research, Lancaster, South Carolina
  - Chattanooga Research & Medicine (CHARM), Chattanooga, Tennessee
  - MultiSpecialty Clinical Research, Inc., Johnson City, Tennessee
  - New Phase Research Development, Knoxville, Tennessee
  - West Houston Clinical Research Services, Houston, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Pulmonary Research of Abingdon, LLC, Abingdon, Virginia
  - TPMG Clinical Research Williamsburg, Williamsburg, Virginia
- Bulgaria (5):
  - SHATPPD - Haskovo, EOOD, Haskovo
  - Medical center Medconsult Pleven OOD, Pleven
  - UMHAT-Plovdiv AD, Plovdiv
  - Medical Center Hera EOOD, Sofia
  - MC "Sv. Ivan Rilski", OOD, Vidin
- Czechia (12):
  - MUDr. I. Cierna Peterova s.r.o., Brandýs nad Labem
  - Fakultni nemocnice Brno, Dept of Klinika nemoci plicnich a tuberkulozy, Brno
  - EDUMED s.r.o., Broumov
  - MUDr. Petr Pravda, Hlučín
  - MediTrial s.r.o., Jindřichův Hradec
  - Plicni ambulance Kralupy s.r.o., Kralupy nad Vltavou
  - CEFISPIRO s.r.o., Lovosice
  - Odborná plicní ambulance Opava s.r.o., Opava
  - DAWON spol. s.r.o., Plicni ambulance, Prague
  - Plicni centrum s.r.o., Prague
  - MUDr. Josef Veverka, Plicni ambulacne, Rokycany
  - Plicni stredisko Teplice s.r.o., Teplice
- Germany (15):
  - MECS GmbH Cottbus, Cottbus, Brandenburg
  - Clinical Studies Pankow Dr Dr Evelin Liefring/Ishak Teber, Berlin, City state Bremen
  - Praxis Dr. Keller, Frankfurt am Main, Hesse
  - IKF Pneumologie GmbH & Co. KG, Frankfurt am Main, Hesse
  - Dr. Christian Schlenska, Peine, Lower Saxony
  - Zentrum fur Klinische Forschung, Cologne, North Rhine-Westphalia
  - Framol-med GmbH, Pneumologische Gemeinschaftspraxis Rheine, Rheine, North Rhine-Westphalia
  - Pneumologische Praxis Dr. Falk Brunner, Leipzig, Saxony
  - Salvus-Klinische Studien GmbH., Leipzig, Saxony
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - PRI Pulmonary Research Institute, Pneumologisches Forschungsinstitut GmbH, Großhansdorf, Schleswig-Holstein
  - KLB Gesundheitsforschung Luebeck GmbH; Praxis Dr. med. Jens Becker, Lübeck, Schleswig-Holstein
  - Studienpraxis Berlin-Brandenburg, Berlin
  - Praxis an der Oper., Berlin
  - Ballenberger, Freytag, Wenisch Institut für klinische Forschung, Neu-Isenburg
- Greece (4):
  - General Hospital of Athens of Chest Diseases "SOTIRIA", 7th Respiratory Clinic, Athens
  - University General Hospital of Heraklion, Pulmonary Clinic, Heraklion
  - University General Hospital of Ioannina, University Respiratory Clinic, Ioannina
  - University General Hospital of Larissa, University Pulmonary Clinic, Larissa
- Hungary (6):
  - Clinexpert Kft., Budapest
  - Szalay János Rendelőintézet Tüdőgyógyászati Szakrendelés, Hajdúnánás
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet Monori Rendelőintézete, Monor
  - Karolina Kórház-Rendelőintézet, Tüdőgyógyászat, Mosonmagyaróvár
  - Püspökladányi Egészségügyi Szolgáltató Nonprofit Kft., Püspökladány
  - Markusovszky Egyetemi Oktatókórház Tüdőgondozó, Szombathely
- Poland (6):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Alergologii Sp. z o. o., Lublin
  - ETG Siedlce, Siedlce
  - NASZ LEKARZ Ośrodek Badań Klinicznych, Torun
  - ETG Warszawa, Warsaw
- Romania (9):
  - S.C Centrul Medical Unirea S.R.L, Campus Medical Brasov, Brasov
  - S.C Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - Spitalul Clinic de Pneumoftiziologie "Leon Daniello" Cluj-Napoca, Brasov
  - Quantum Medical Center S.R.L., Bucharest
  - Institutul de Pneumoftiziologie "Marius Nasta", Bucharest
  - S.C Cardiomed S.R.L, Cluj-Napoca
  - Impatiens SRL, Codlea
  - Fundatia Cardioprevent, Timișoara
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie "Dr. Victor Babes" Timisoara, Timișoara
- Russia (16):
  - NSHI "Departmental CH on St. Barnaul of JSCO "Russian Railways", Barnaul
  - SBHI "Regional Clinical Hospital #3", Chelyabinsk
  - FSBI "Scientific-research Institute for Complex Problems of cardiovascular disease", Kemerovo
  - LLC "Novosibirsk GastroCenter", Novosibirsk
  - SBIH of Novosibirsk Region "Clinical Emergency Hospital #2", Novosibirsk
  - City Clinical Hospital #25, Novosibirsk
  - SPb SBHI "Vvedenskaya hospital", Saint Petersburg
  - "LEC at the LLC "LLC "Energiy Zdorovya", Saint Petersburg
  - LLC "Institute of Medical Examinations", Saint Petersburg
  - Research center Eco-safety, LLC, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
  - SBHI of Yaroslavl Region "Clinical Hospital # 2", Yaroslavl
  - SBHI Outpatient 2, Yaroslavl
  - LLC MA New Hospital, Yekaterinburg
  - City Hospital #6, Yekaterinburg
- Slovakia (3):
  - Nemocnica s poliklinikou Sv. Jakuba, n.o. Bardejov, Bardejov
  - Inspiro, s.r.o., Humenné
  - Plucna ambulancia Hrebenar, s.r.o., Spišská Nová Ves
- South Korea (5):
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
- Respiratory Clinical Trials Ltd, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Dransfield M, Marchetti N, Kalhan R, Reyner D, Dixon AL, Rheault T, Rickard KA, Anzueto A. Ensifentrine in COPD patients taking long-acting bronchodilators: A pooled post-hoc analysis of the ENHANCE-1/2 studies. Chron Respir Dis. 2025 Jan-Dec;22:14799731251314874. doi: 10.1177/14799731251314874. PMID 39854278
- [Derived] Sciurba FC, Christenson SA, Rheault T, Bengtsson T, Rickard K, Barjaktarevic IZ. Effect of Dual Phosphodiesterase 3 and 4 Inhibitor Ensifentrine on Exacerbation Rate and Risk in Patients With Moderate to Severe COPD. Chest. 2025 Feb;167(2):425-435. doi: 10.1016/j.chest.2024.07.168. Epub 2024 Aug 27. PMID 39197510
- [Derived] Mahler DA, Bhatt SP, Rheault T, Reyner D, Bengtsson T, Dixon A, Rickard K, Singh D. Effect of ensifentrine on dyspnea in patients with moderate-to-severe chronic obstructive pulmonary disease: pooled analysis of the ENHANCE trials. Expert Rev Respir Med. 2024 Aug;18(8):645-654. doi: 10.1080/17476348.2024.2389960. Epub 2024 Aug 8. PMID 39106052
- [Derived] Anzueto A, Barjaktarevic IZ, Siler TM, Rheault T, Bengtsson T, Rickard K, Sciurba F. Ensifentrine, a Novel Phosphodiesterase 3 and 4 Inhibitor for the Treatment of Chronic Obstructive Pulmonary Disease: Randomized, Double-Blind, Placebo-controlled, Multicenter Phase III Trials (the ENHANCE Trials). Am J Respir Crit Care Med. 2023 Aug 15;208(4):406-416. doi: 10.1164/rccm.202306-0944OC. PMID 37364283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, randomized, double-blind, placebo-controlled study was conducted in patients with moderate to severe chronic obstructive pulmonary disease (COPD) at 120 study centers in 12 countries between 29 Sep 2020 and 02 Dec 2022. Patients were randomized in a 5:3 ratio overall (1:1 over 24 weeks and 3:1 over 48 weeks), stratified by duration, smoking status and background medication use, to receive either ensifentrine or placebo.
Pre-assignment Details: Patients were screened for eligibility before entering a 28-day run in period to ensure a stable COPD treatment regimen and to collect baseline information on symptoms and rescue medication use.
Groups:
- Ensifentrine: 3 milligram (mg) twice daily via standard jet nebulizer.
- Placebo: Twice daily via standard jet nebulizer.
Period: Overall Study
Arm/Group | Ensifentrine | Placebo
Started | 479 | 284
Received Treatment | 477 | 283
Completed | 400 | 245
Not Completed | 79 | 39
Not completed — Death | 4 | 5
Not completed — COPD exacerbation withdrawal criteria | 7 | 5
Not completed — Coronavirus disease 2019 (COVID-19) | 8 | 6
Not completed — Adverse Event | 10 | 1
Not completed — Lack of Efficacy | 3 | 2
Not completed — Investigator discretion | 3 | 0
Not completed — Withdrawal by Subject | 32 | 14
Not completed — Lost to Follow-up | 5 | 3
Not completed — Other | 7 | 3

BASELINE CHARACTERISTICS:
Population: All patients randomized set included all patients in the enrolled set who were randomized to study medication.
Groups:
- Ensifentrine: 3 mg twice daily via standard jet nebulizer.
- Total: Total of all reporting groups
Arm/Group | Ensifentrine | Placebo | Total
Number analyzed (Participants) | 479 | 284 | 763
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.12) | 64.9 (7.73) | 65.0 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 117 | 321
  Male | 275 | 167 | 442
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 11 | 24
  Black or African American | 16 | 9 | 25
  White | 437 | 251 | 688
  Other | 0 | 1 | 1
  Not Reported | 13 | 12 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 6 | 21
  Not Hispanic or Latino | 464 | 278 | 742
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 28 | 17 | 45
  Czechia | 70 | 36 | 106
  Germany | 117 | 73 | 190
  Greece | 3 | 3 | 6
  Hungary | 25 | 14 | 39
  South Korea | 12 | 11 | 23
  Poland | 10 | 3 | 13
  Romania | 21 | 18 | 39
  Russia | 71 | 33 | 104
  Slovakia | 27 | 14 | 41
  United Kingdom | 8 | 4 | 12
  United States | 87 | 58 | 145

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline in Average Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve Over 12 Hours (AUC0-12h) at Week 12
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Average FEV1 AUC0-12h was defined as AUC over 12 hours of the FEV1, divided by 12 hours. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on Day 1. Spirometry assessments were performed in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines.
Time Frame: Baseline (pre-dose on Day 1) and Week 12
Population: The modified Intent-to-Treat (mITT) population set included all patients in the randomized set who received at least 1 dose (or partial dose) of study medication, and patients were classified according to randomized treatment. 1 patient was missing a baseline FEV1 assessment.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 477 | 282
liters | 0.0611 (0.01825) | -0.0256 (0.0195)
Statistical Analysis 1: Comparison: Ensifentrine vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The analysis of covariance (ANCOVA) model was used to model the change from baseline FEV1 to average FEV1 AUC0-12h with treatment, region, background medication strata and smoking strata as fixed effects and baseline FEV1 as covariate; LS mean difference = 0.0868, 95% CI 2-sided [0.0551 to 0.1185], Standard Error of Mean 0.0162

2. Secondary Outcome: LS Mean Change From Baseline FEV1 to Peak FEV1 at Day 1 and Weeks 6, 12 and 24
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Peak FEV1 is the maximum value in the 4 hours after dosing. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on Day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (pre-dose on Day 1), post-dose on Day 1, Weeks 6, 12, and 24
Population: The mITT population set included all patients in the randomized set who received at least 1 dose (or partial dose) of study medication, and patients were classified according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 477 | 282
liters
  Day 1 (Post-dose) | 0.2274 (0.0130) | 0.0755 (0.0138)
  Week 6 | 0.2038 (0.0193) | 0.0677 (0.0207)
  Week 12 | 0.2042 (0.0201) | 0.0570 (0.0217)
  Week 24 | 0.1623 (0.0217) | 0.0462 (0.0234)

3. Secondary Outcome: LS Mean Change From Baseline to the Mean Weekly Evaluating-Respiratory Symptoms (E-RS) Total Score at Weeks 6, 12 and 24
Description: The E-RS scale consists of 11 questions, with 3 sub-domains of: breathlessness, cough and sputum, and chest symptoms. The E-RS sub-domain score was calculated as the sum from the relevant questions. The E-RS total score was derived as the sum of the raw scores of the 11 items ranging from 0 to 40. Higher scores indicates severe respiratory symptoms. Scores were derived weekly as the mean over 7 days prior to the visit, using only days where data was recorded. The E-RS was collected daily by electronic diary (e-diary). Baseline is the mean over the 7 days prior to the first intake of study medication, using only days where data was recorded.
Time Frame: Baseline (pre-dose on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 475 | 281
units on a scale
  Week 6 | -1.944 (0.3581) | -1.157 (0.3831)
  Week 12 | -2.498 (0.3897) | -1.127 (0.4176)
  Week 24 | -2.249 (0.4247) | -1.298 (0.4573)

4. Secondary Outcome: LS Mean Change From Baseline in the St. George's Respiratory Questionnaire (SGRQ) Total Score at Weeks 6, 12 and 24
Description: The SGRQ questionnaire consists of 17 questions, split into 2 parts. Part 1 consisted of the first 8 questions and was related to the symptoms subdomain. The remaining 9 questions were in Part 2, which were related to the activity and impacts subdomains. The total score was calculated by dividing the summed weights by the maximum possible weight for all items in the questionnaire and expressing the result as a percentage. Score ranging from 0 to 100 and higher scores indicated a worse outcome. Baseline is the score calculated on Day 1 prior to 4 hour post-dose spirometry.
Time Frame: Baseline (pre-dose on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 474 | 281
units on a scale
  Week 6 | -6.184 (0.9838) | -3.965 (1.0511)
  Week 12 | -5.665 (1.0163) | -2.652 (1.0859)
  Week 24 | -6.167 (1.1405) | -3.868 (1.2178)

5. Secondary Outcome: LS Mean Change From Baseline FEV1 to Morning Trough FEV1 at Weeks 6, 12 and 24
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Morning trough FEV1 was the last value collected prior to the morning dose. Baseline FEV1 is the mean of the two measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (pre-dose on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 477 | 282
liters
  Week 6 | 0.0112 (0.0181) | -0.0259 (0.0193)
  Week 12 | 0.0076 (0.0190) | -0.0272 (0.0204)
  Week 24 | -0.0236 (0.0205) | -0.0369 (0.0219)

6. Secondary Outcome: LS Mean Change From Baseline in Average FEV1 Area Under the Curve Over 4 Hours (AUC0-4h) at Day 1 and Weeks 6, 12 and 24
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Average FEV1 AUC0-4h was defined as area under the curve over 4 hours of the FEV1, divided by 4 hours. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on Day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (pre-dose on Day 1), post-dose on Day 1, Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 477 | 282
liters
  Day 1 (Post-dose) | 0.1495 (0.0108) | 0.0099 (0.0115)
  Week 6 | 0.1259 (0.0184) | -0.0044 (0.0196)
  Week 12 | 0.1243 (0.0191) | -0.0149 (0.0203)
  Week 24 | 0.0875 (0.0206) | -0.0139 (0.0220)

7. Secondary Outcome: Percentage of SGRQ Responders at Weeks 6, 12 and 24
Description: The SGRQ questionnaire consists of 17 questions, split into 2 parts. Part 1 consisted of the first 8 questions and was related to the symptoms subdomain. The remaining 9 questions were in Part 2, which were related to the activity and impacts subdomains. The total score was calculated by dividing the summed weights by the maximum possible weight for all items in the questionnaire and expressing the result as a percentage. Responder was a patient with an improvement from baseline in SGRQ total score of 4 or more. Percentage of SGRQ responders are reported.
Time Frame: Weeks 6, 12 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 474 | 281
percentage of patients
  Week 6 | 50.8 | 40.6
  Week 12 | 52.5 | 37.0
  Week 24 | 58.2 | 45.9

8. Secondary Outcome: LS Mean Change From Baseline to the Mean Weekly Rescue Medication Use at Weeks 6, 12 and 24
Description: Use of rescue medication (albuterol/salbutamol) per week was calculated as the LS mean use daily over 7 days. Daily rescue medication use was collected in an e-diary throughout the study. Baseline is the mean over the 7 days prior to the first intake of study medication, calculated as the sum of puffs taken, divided by number of days data has been recorded.
Time Frame: Baseline (pre-dose on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: rescue medication puffs per week
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 475 | 281
rescue medication puffs per week
  Week 6 | -0.442 (0.1065) | -0.306 (0.1139)
  Week 12 | -0.469 (0.1155) | -0.182 (0.1234)
  Week 24 | -0.506 (0.1448) | -0.052 (0.1554)

9. Secondary Outcome: LS Mean Transition Dyspnea Index (TDI) Questionnaire Total Score at Weeks 6, 12 and 24
Description: The TDI is a questionnaire that focused on 3 sub-domains: functional impairment, magnitude of task and magnitude of effort. Sub-domain score was calculated as the sum from the related questions. Total score was calculated as the sum of the sub-domain scores. The TDI measures the change in dyspnea severity from the baseline as measured by the baseline dyspnea index. It was rated by 7 grades ranging from -3 (major deterioration) to +3 (major improvement). Higher scores indicate better outcome. Change from baseline was assessed with the Baseline Dyspnea Index.
Time Frame: Weeks 6, 12 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 471 | 277
units on a scale
  Week 6 | 1.3 (0.19) | 0.6 (0.21)
  Week 12 | 1.6 (0.21) | 0.4 (0.23)
  Week 24 | 1.9 (0.24) | 0.8 (0.27)

10. Secondary Outcome: LS Mean Change From Baseline FEV1 to Evening Trough FEV1 at Week 12
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Evening trough FEV1 was the value collected at 12 hours post-morning dose and prior to the evening dose. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (pre-dose on Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 477 | 282
liters | -0.0117 (0.0203) | -0.0697 (0.0214)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs; serious or non-serious), were collected from first dose of study medication up to 10 days after final study visit (24-week subset: at Week 24, approximately 25 weeks; 48-week subset: at Week 48, approximately 49 weeks). Serious Adverse Events (SAEs) assessed as related to study participation (eg, change in existing therapy) and which occurred prior to first dose of study medication were collected from time of consent through follow-up contact.
Description: The safety analysis included all randomized patients who received at least 1 dose (or partial dose) of study medication. TEAEs (serious or non-serious) that started or worsened in severity on or after first dose of study medication are reported. SAEs assessed as related to study participation and which occurred prior to first dose of study medication are not reported as it was pre-specified to report only TEAEs that started or worsened in severity on or after first dose of study medication.
Groups:
- Up to Week 24: Ensifentrine: 3 mg twice daily via standard jet nebulizer.
- Up to Week 24: Placebo: Twice daily via standard jet nebulizer.
- From Week 24 to Week 48: Ensifentrine: 3 mg twice daily via standard jet nebulizer (patients that had at least 1 dose after Week 24 visit).
- From Week 24 to Week 48: Placebo: Twice daily via standard jet nebulizer (patients that had at least 1 dose after Week 24 visit).
Arm/Group | Up to Week 24: Ensifentrine | Up to Week 24: Placebo | From Week 24 to Week 48: Ensifentrine | From Week 24 to Week 48: Placebo
All-Cause Mortality (participants affected / at risk) | 2/477 | 4/283 | 2/228 | 1/70
Serious Adverse Events (participants affected / at risk) | 32/477 | 19/283 | 11/228 | 5/70
Other Adverse Events (participants affected / at risk) | 90/477 | 58/283 | 16/228 | 17/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Up to Week 24: Ensifentrine (N=477) | Up to Week 24: Placebo (N=283) | From Week 24 to Week 48: Ensifentrine (N=228) | From Week 24 to Week 48: Placebo (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 2 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 3 | 1 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 1
Myocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pharyngeal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral microangiopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Up to Week 24: Ensifentrine (N=477) | Up to Week 24: Placebo (N=283) | From Week 24 to Week 48: Ensifentrine (N=228) | From Week 24 to Week 48: Placebo (N=70)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 6 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 16 | 9 | 2 | 2
Cellulitis (Infections and infestations) | 0 | 3 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 13 | 16 | 6 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 4 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 4 | 0 | 0
Headache (Nervous system disorders) | 16 | 12 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 11 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT04535986/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT04535986/SAP_001.pdf